CLINICAL TRIAL: NCT05039060
Title: A Modified Microbiota-Accessible Carbohydrates (MAC) Diet and Change of Gut Microbiota in Patients With Colorectal Cancer After Surgery: A Prospective, Open-label, Cross-over, Single Center Study
Brief Title: Modified MAC Diet and Gut Microbiota in CRC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: modifiedMAC001
Record Dates: First submitted 2021-08-10; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer; Gut Microbiota; Diet Intervention
Keywords: Colorectal Cancer; Gut Microbiota; microbiota accessible carbohydrates
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Approximately 40 participants will be randomly assigned to following group (group 1 or group 2). The subjects will be consumed the modified MAC or conventional diet for first 3-weeks period then cross-over to second 3-weeks period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1: Modified MAC diet (first 3-weeks) followed by conventional diet (second 3-weeks)
  Interventions: Dietary Supplement: Modified MAC diet (3-weeks)
- Group 2 (Placebo Comparator): Group 2: Conventional diet (first 3-weeks) followed by modified MAC diet (second 3-weeks)
  Interventions: Dietary Supplement: Modified MAC diet (3-weeks)

INTERVENTIONS:
Dietary Supplement: Modified MAC diet (3-weeks) — * Modified MAC diet to adapt reduced energy intake and increased dietary fiber consumption with appropriate nutrients component
  * Dr.Kitchen Inc. directly provide home delivery service for the modified MAC diet including multigrain rice, meal kit, and snacks per day in a regular basis

SUMMARY:
To explore the changes in the composition and diversity of intestinal microbiota during 3-weeks of modified MAC diet and conventional diet in stage I or low-risk stage II colorectal cancer (CRC) patients after surgery. Additionally, the investigator analyze the association of gut microbiota and stool formation pattern or quality of life according to dietary pattern. Therefore, the investigator identify the beneficial or harmful microbiota composition and diversity adapting modified MAC diet that related to cancer recurrence, which provide supporting evidence for future prospective trial.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer worldwide and a life-threatening disease that kills more than 500,000 people every year. It is known that, environmental factors such as diet and lifestyle play an important role in the development of colorectal cancer due to large differences in the incidence rate by region in addition to the genetic background associated with colorectal cancer. The physical activity, whole grains, dietary fiber, dairy products, and calcium supplement intake are factors that inhibit colorectal cancer, but red meat, processed meat, alcohol, and obesity act as risk factors inducing colorectal cancer. Therefore, it can be said that efforts to prevent cancer are important compared to other cancers.

A growing interest in the interaction of the gut microbiome with its host and its important role in health and disease is revealing that the interaction of the gut microbiome with humans plays an important role in the development of degenerative diseases, cancers and inflammatory diseases. According to recent studies, the risk of colorectal cancer is increased by the presence of specific gut microbiota, dysbiosis, and the interaction between diet and gut microbes. In other words, changes in diet affect the formation of the intestinal microbiota, and conversely, microorganisms mediate the generation of dietary factors that cause colorectal cancer.

In addition, microorganisms such as Fusobacterium nucleatum regulate autophagy and play a role in making it resistant to chemotherapy after colon cancer surgery, or whole grains in colorectal cancer patients with Fusobacterium nucleatum in tumor tissue. However, a cohort study has also reported that consuming a diet rich in dietary fiber helps to lower the incidence of colorectal cancer.

Diet and nutrients play a decisive role in the composition of the intestinal microflora involved in the regulation of inflammation and immune responses.

Microbiota-Accessible Carbohydrates (MAC) refer to carbohydrates that the human intestine cannot digest, but that can be digested by intestinal microbes. It is not decomposed and not absorbed in the stomach or small intestine, and then broken down in the large intestine and then digested and metabolized by the intestinal microflora. During that process, short chain fatty acid (SCFA) is produced, which is known to increase beneficial intestinal bacteria and decrease inflammation around intestinal cells.

The composition of intestinal microbes changes due to intestinal preparation before colon cancer surgery, use of prophylactic antibiotics, and tissue changes in the intestine anastomosis, which may lead to enhanced toxicity, proliferation of pathogens, and reduction of beneficial intestinal bacteria. In addition, the presence of certain microorganisms may lead to complications such as anastomotic leakage or infection at the surgical site.

Thanks to the development of various genomic research techniques, there is a difference in the composition of intestinal microbes between colorectal cancer patients and healthy people, and the microbiome affects the development of adenoma or cancer as the number of beneficial bacteria decreases, the harmful bacteria changes in terms of age.

In this study, a modified MAC diet designed to adapt to a high-fiber diet after surgery and a patient-made diet for stage 1-2 colorectal cancer patients who do not receive chemotherapy after colon cancer surgery using the genomic analysis technique The purpose of this study is to explore the effect of diet on the composition of the intestinal microflora, and to analyze whether the different diet affects the pattern of defecation after colorectal cancer surgery, and the effect of these changes on the quality of life after colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed colorectal adenocarcinoma patients after curative surgery without post-operative chemotherapy (stage I and low-risk stage II)
2. Male of female participants over the age of 19
3. Eastern Cooperative Oncology Group (ECOG) performance score 0-2
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol
5. Adequate hematologic and end-organ function

Exclusion Criteria:

1. Patients with temporary/permanent stoma after surgery
2. Diagnosed with locally advanced stage (more than high-risk stage II) colorectal cancer which require postoperative chemotherapy after surgery
3. Diagnosed with metastatic stage IV colorectal cancer after surgery
4. Uncontrolled diabetes (glycated hemoglobin A1c (HbA1c) > 8.0 g/dl)
5. Active infection requiring antibiotics, antifungal or antiviral agents or received a course of antibiotics within 4 weeks prior to study treatments
6. Known history of food allergy
7. Known history of uncontrolled intercurrent illness including but not limited to: Infection/inflammation; severe liver dysfunction; bilateral interstitial lung disease; uncontrolled kidney disease; clinically significant (active) cardiovascular and pulmonary disease; hemorrhagic disease; inflammatory bowel disease, intestinal obstruction; Inability to swallow food; social and psychological problems etc.)
8. Other medical and psychiatric conditions that would prohibit the understanding or rendering of informed consent which affect study compliance

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
The change of gut microbiota diversity | Stool sample collection for baseline, after the first 3-week diet, and then after second 3-week diet
  a-diversity for interpersonal change and b-diversity for groups using 16s rRNA sequencing

SECONDARY OUTCOMES:
The change of stool formation pattern | Up to 6 week (during study period)
  Daily check for stool pattern using Bristol Stool Score
The change of quality of life | Survey for baseline, after the first 3-week diet, and then after second 3-week diet
  3 times check for quality of life using EORTC QLQ-C30 plus QLQ-CR29 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire 30 items for Common function and symptom plus 29 items specific for colorectal cancer, It is converted into a score range from 0-100, and the overall quality of life score is high, The higher the functional domain score and the lower the symptom domain score, the better the quality of life.)
The change of quality of life | Survey for baseline, after the first 3-week diet, and then after second 3-week diet
  3 times check for quality of life using EORTC QLQ-C30 plus QLQ-CR29
The change of gut microbiota metabolite | Stool sample collection for baseline, after the first 3-week diet, and then after second 3-week diet
  Analysis for gut microbiota producing short chain fatty acid

CONTACTS AND LOCATIONS:
Overall Officials: Soohyeon Lee, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No